CLINICAL TRIAL: NCT05652556
Title: Quinolone Resistance Profiles and Mechanisms of Staphylococcus Aureus and Escherichia Coli From Humans, Chicken and Catfish Farms With a One Health Approach in Blitar, East Java Province, Indonesia
Brief Title: Quinolone Resistance Profiles and Mechanisms of Staphylococcus Aureus and Escherichia Coli From Humans, Chicken and Catfish Farms in Indonesia
Acronym: QUINDO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dr. Soetomo General Hospital (Other Government); Balai Besar Laboratorium Kesehatan (BBLK) Surabaya (Unknown); National Institute of Health Research and Development, Ministry of Health Republic of Indonesia (Other); Directorate of Veterinary Public Health, Ministry of Agriculture, Indonesia (Unknown); Directorate of Animal Health, Ministry of Agriculture, Indonesia (Unknown); Ministry of Marine and Fisheries, Indonesia (Unknown); Utrecht University (Other); Radboud University Medical Center (Other); National Institute for Public Health and the Environment (RIVM) (Other Government)
Responsible Party: Principal Investigator, Juliëtte Severin, Associate professor, Medical coordinator Unit infection prevention, Erasmus Medical Center
Other Study IDs: QUINDO
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Drug Resistance, Microbial
Keywords: Escherichia coli; Staphylococcus aureus; Fluoroquinolones
MeSH Terms: conditions — Escherichia coli Infections; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Culture of nasal and rectal swabs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to reveal quinolone resistance profiles and mechanisms in S. aureus and E. coli in the human, animal and aquaculture sector in Blitar, Indonesia.

The main questions it aims to answer are:

* Obtain the quinolone resistance profiles and mechanisms of S. aureus and E. coli in human health, animal health and aquaculture health sector in Blitar, Indonesia.
* Obtain the association of AMR and AMU data within and between the human health, animal health and aquaculture health sector in Blitar, for quinolones.

DETAILED DESCRIPTION:
Antimicrobial resistance (AMR) has become a global threat in public health. It is mainly driven by antimicrobial use (AMU), not only in the human sector, but also in the animal and aquaculture sector. In aquaculture and terrestrial animals, antibiotics have been used as growth promoters as well as for prophylaxis and treatment for infection. It has been used on a large scale as a supplement to increase animal production in over 60 years. During the last decade, there has been an increasing antimicrobial resistance in the community regarding resistance to carbapenems, 3rd generation cephalosporins and quinolones. The World Health Organization categorized carbapenems, 3rd generation cephalosporins and quinolones as "Watch antibiotics" and these should be used with caution because of their high effects and their high potential to cause the development of AMR in many countries.

The quinolones are broad-spectrum antibiotics that are probably one of the most widely used drugs for the treatment of several community and hospital-acquired infections in the human health sector. It is also used in aquaculture and agricultural fields, for instance in chicken farms. The use of quinolones and other "Watch antibiotics" in many countries monitored by the World Health Organization since 2016 varies a lot and ranges from less than 20% to more than 50%.

It is well documented that several pathogenic bacteria have developed resistance as a consequence of exposure to the antimicrobials. Resistant bacteria can spread to humans directly from the food chain, and indirectly from the environmental pollution of farm effluents. This study will reveal quinolone resistance profiles and mechanisms in S. aureus and E. coli in the human, animal and aquaculture sector in Blitar, Indonesia.

Population The research populations are residents (farmers and non-farmers) in Kabupaten Blitar.

Sample

Layer farm:

Samples will be taken in layer farms in the Blitar region. The type of sample will be bootswab samples as published before; 25 E. coli isolates/farm will be collected. A total of 30 farms will be included.

Aquaculture sample:

Aquaculture samples will be taken from catfish ponds in several regions in Kabupaten Blitar. One sample of water or mud of one pond will be taken (the pond closest to the entrance). From this sample, 5 E. coli will be isolated.

Human sample:

Human samples will be taken from people on layer and aquaculture farms (farmers, farmworkers and family members of farmers), and non-farmer residents of several regions in Kabupaten Blitar. Nasal (S. aureus) and rectal (E. coli) samples will be taken after informed consent. AMU data will be collected via questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Farmers of included farms and non-farmers. Non-farmers will be approached via public health center (puskesmas).
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2022-12-09 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Quinolone resistance profiles and mechanisms of S. aureus and E. coli in human health, animal health and aquaculture health sector in Blitar | 2023
  As determined by Vitek, microdilution, and whole genome sequencing.

SECONDARY OUTCOMES:
Association of AMR and AMU data within and between the human health, animal health and aquaculture health sector in Blitar, for quinolones | 2023
  Based on questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Juliëtte A. Severin, MD PhD, Principal Investigator — Erasmus Medical Center

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet.